CLINICAL TRIAL: NCT02060929
Title: An Open-Label Phase 1 Study to Evaluate the Pharmacokinetics of Intranasal Esketamine Administered With and Without a Nasal Guide on the Intranasal Device
Brief Title: A Study to Evaluate the Pharmacokinetics of Intranasal Esketamine Administered With and Without a Nasal Guide on the Intranasal Device
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR102971; ESKETINTRD1004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-01-21; First posted 2014-02-12 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: Healthy; Esketamine; Intranasal; Nasal Guide; Pharmacokinetics
MeSH Terms: interventions — Esketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): Participants will self administer 1 spray of esketamine solution to each nostril using a intranasal (through nose) device with a nasal guide on Day 1 of period 1 as treatment regimen A at time 0 and repeated twice every 5 minutes (total dose: 84 mg). There will be a washout period of 5-10 days between the treatment regimens. On Day 1 of period 2, participants will self administer 1 spray of esketamine solution to each nostril using a intranasal device without a nasal guide as treatment regimen B at time 0 and repeated twice every 5 minutes (total dose: 84 mg).
  Interventions: Drug: Esketamine
- Sequence 2 (Experimental): Participants will self administer 1 spray of esketamine solution to each nostril using a intranasal device without a nasal guide on Day 1 of period 1 as treatment regimen B at time 0 and repeated twice every 5 minutes (total dose: 84 mg). There will be a washout period of 5-10 days between the treatment regimens. On Day 1 of period 2, participants will self administer 1 spray of esketamine solution to each nostril using a intranasal device with a nasal guide as treatment regimen A at time 0 and repeated twice every 5 minutes (total dose: 84 mg).
  Interventions: Drug: Esketamine

INTERVENTIONS:
Drug: Esketamine — Participants will self administer 1 spray of esketamine solution using a intranasal device with a nasal guide in Treatment A regimen and without nasal guide inTreatment B regimen at time 0 and repeated twice every 5 minutes (total dose: 84 mg).

SUMMARY:
The primary purpose of the study is to evaluate the pharmacokinetics (what the body does to the medication) of intranasally (through the nose) administered esketamine using a device with and without a nasal guide in healthy participants.

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by chance), single-center, single-dose, 2-way crossover (participants may receive different interventions sequentially during the study in 2 sequence groups), open-label (all people know the identity of the intervention) study. Approximately, 14 participants will be enrolled in this study. This study will consist of a screening phase of up to 21 days, a treatment phase of 3 days, and a follow-up phase of 9-13 days. Participants will be randomly allocated to 1 of the 2 treatment groups (Sequence 1 and 2). In sequence 1, participants will self-administer esketamine intranasally using a device with nasal guide as treatment A on Day 1 of period 1 and intranasally esketamine using a device without nasal guide as treatment B on Day 1 of period 2. In sequence 2, participants will self-administer intranasally esketamine as treatment B on Day 1 of period 1 and intranasally esketamine as treatment A on Day 1 of period 2. There will be a washout period of 5 to 10 days between each treatment regimen. Safety evaluations will include assessment of adverse events, clinical laboratory tests, electrocardiogram, vital signs, physical examination, pulse oximetry, targeted nasal examination, nasal device questionnaire, and in addition to these evaluations, specific scales will be used to assess the safety. The study duration for each participant will be approximately 45 days.

ELIGIBILITY:
Inclusion Criteria:

* Agrees to protocol-defined use of effective contraception
* If a woman, must have a negative serum human chorionic gonadotropin (hCG) pregnancy test at screening; and a negative urine pregnancy test on Day -1 of each treatment period
* Body mass index (BMI) (weight [kg]/height2 [m]2) between 18 and 30 kg/m2 (inclusive), and body weight not less than 50 kg
* Blood pressure (after the participant is supine for 5 minutes) between 90 and 140 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic
* A 12-lead electrocardiogram (ECG) consistent with normal cardiac conduction and function

Exclusion Criteria:

* Current or prior history of psychiatric disorder including but not limited to psychotic, bipolar, major depressive, or anxiety disorder
* Clinically significant medical illness including cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders , lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic disease, infection, hypertension or vascular disorders, kidney or urinary tract disturbances, sleep apnea, myasthenia gravis, or any other illness
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening or at admission to the study center (Day -1) as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs, or 12-lead ECG at screening or at admission to the study center (Day -1 of each treatment period) as deemed appropriate by the investigator
* Has an abnormal or deviated nasal septum with any 1 or more of the following symptoms: blockage of 1 or both nostrils, nasal congestion (especially 1-sided), frequent nosebleeds, frequent sinus infections, noisy breathing during sleep, facial pain, headaches, and postnasal drip

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Esketamine | Pre-dose, and post-dose 7, 12, 22, 32, 40, 50 minutes, 1, 1.25, 1.5, 2, 3, 4, 24 hours
  Cmax is defined as maximum observed analyte concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of Esketamine | Pre-dose, and post-dose 7, 12, 22, 32, 40, 50 minutes, 1, 1.25, 1.5, 2, 3, 4, 24 hours
  Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Time at Last Observed Quantifiable Concentration (AUClast) of Esketamine | Pre-dose, and post-dose 7, 12, 22, 32, 40, 50 minutes, 1, 1.25, 1.5, 2, 3, 4, 24 hours
  The AUClast is area under the plasma concentration-time curve from time zero to the last quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of Esketamine | Pre-dose, and post-dose 7, 12, 22, 32, 40, 50 minutes, 1, 1.25, 1.5, 2, 3, 4, 24 hours
  The AUC(0-infinity) is area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of Area under Curve (AUC) last and C(last)/lambda(z), in which C(last) is the last observed quantifiable concentration
Elimination Half-Life Period (T1/2) of Esketamine | Pre-dose, and post-dose 7, 12, 22, 32, 40, 50 minutes, 1, 1.25, 1.5, 2, 3, 4, 24 hours
  T1/2 is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal rate-constant (lambda[z]) of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
First-order Rate Constant of Esketamine | Pre-dose, and post-dose 7, 12, 22, 32, 40, 50 minutes, 1, 1.25, 1.5, 2, 3, 4, 24 hours
  First-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Relative Bioavailability (Frel) of Esketamine | Pre-dose, and post-dose 7, 12, 22, 32, 40, 50 minutes, 1, 1.25, 1.5, 2, 3, 4, 24 hours
  Relative bioavailability is the percentage of the administered dose that is systemically available.
Change From Baseline in Clinician-Administered Dissociative States Scale (CADSS) Score | Baseline (Day -1) and Day 2
  The CADSS is a clinician administered rating scale designed to measure dissociative symptoms. The CADSS comprises 23 subjective items, divided into 3 components: depersonalization, derealization and amnesia. Participant's responses are coded on a 5-point scale (0 = "Not at all" through to 4 = "Extremely). Higher scores indicate worsening.
Change From Baseline in Brief Psychiatric Rating Scale (BPRS) Score | Baseline (Day -1) and Day 2
  The BPRS is used for the measurement of psychiatric symptoms. The BPRS is an 18 item questionnaire and each question is rated on a 7-point scale ranging from 1 (not present) to 7 (extremely severe). The total score for the 18 question will be calculated by adding score of each question. The interpretation of the total scores are: 0-9 will indicate "not a schizoaffective case"; 10-20 will indicate "possible schizoaffective case"; and 21 or more, will indicate "evident schizoaffective case". Higher scores indicate worsening.
Change From Baseline in Modified Observers Assessment of Alertness/Sedation (MOAA/S) Score | Baseline (Day 1) and Day 2
  The MOAA/S is a 6-point ordinal scale measuring a patient's level of sedation. Scores range from 0 (No response to painful stimulus [trapezius squeeze]) to 5 (Responds readily to name spoken in normal tone [awake]). MOAA/S scores were classified as 0-1, 2-4 and 5.
Change From Baseline in Columbia Suicide Severity Rating Scale (C-SSRS) Score | Baseline (Screening - Day -21 to Day -2) and follow-up visit (11 to 13 days after final dose)
  The C-SSRS is a clinical interview to assess severity and track suicidal events providing a summary of both suicidal ideation and behavior to identify the level and type of suicidality present.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium